CLINICAL TRIAL: NCT05063422
Title: Retentive Strength of Various Dental Adhesives on Various Types of Residual Ridged
Brief Title: Retentive Strength of Denture Adhesives on Various RR Ridges
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Altamash Institute of Dental Medicine (Other)
Responsible Party: Principal Investigator, Dr Maria Shakoor, Asistant Professor (BDS, FCPS), Altamash Institute of Dental Medicine
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Supportive Care
Other Study IDs: Denture adhesive
Record Dates: First submitted 2021-06-24; First posted 2021-10-01 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Retentive Strength of Denture Adhesives
Keywords: alveolar ridge resorption; denture adhesives
MeSH Terms: interventions — Carboxymethylcellulose Sodium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Mild Resorption of mandibular ridge (Experimental): Loss of upto 1/3 of original vertical height
  Interventions: Drug: polymyxin b/trimethoprim ophthalmic, Carboxymethyl cellulose
- Moderate Resorption of mandibular ridge (Experimental): 2. Moderate Resorption: Loss of upto 1/3 to 2/3 of original vertical height
  Interventions: Drug: polymyxin b/trimethoprim ophthalmic, Carboxymethyl cellulose
- Severe Resorption of mandibular ridge (Experimental): 3. Severe Resorption: Loss of 2/3 or more of original vertical height
  Interventions: Drug: polymyxin b/trimethoprim ophthalmic, Carboxymethyl cellulose

INTERVENTIONS:
Drug: polymyxin b/trimethoprim ophthalmic, Carboxymethyl cellulose — 3 forms of denture adhesives from each brands are used to compare the retentive strength on highly resorbed ridges

SUMMARY:
To compare the retentive strength of different form of commercially available denture adhesives (paste, powder and cushion) on different form of residual ridges.

To evaluate the effect of various denture adhesives on efficiency of complete dentures in patients with different alveolar ridges.

DETAILED DESCRIPTION:
* Prior approval from ethical committee has been taken (Annexure-D)
* As per protocol all patients presenting will be examined in general opd and those patients in need of rehabilitation of their missing teeth will be referred to Prosthodontics dept.
* Patients will undergo history and complete oral examination after informed consent (Annexure-B). On the basis of these information the patient will be selected for the study acc to exclusion and inclusion criteria.
* The patients will then categorized into three groups based on clinical and radiographic features of ridges according to Wical-Swoope classification.
* A well-constructed denture will be fabricated and all the post op complaints will be resolved.
* Three forms of denture adhesives will be used including powder, cream and strips for all three resorption classes as described by Wical-Swoope.
* A digital spring scale will be used to record the reading , All the measurements will be recorded in grams
* Retentive strength will be recorded first before application of the adhesives for baseline retention strength.
* Patient with denture in his mouth will be instructed to maintain max non-forced intercuspation for fives minutes. Atfer that with mouth opened and lower lip relaxed in order to avoid losing peripheral seal tip of the spring scale will be placed at the margin of denture in recess to lingual frenum. Traction forced will be then applied until denture is detached, the max retention force being recorded by sping scale. This procedure will be repeated thrice and mean value will be calculated.
* A second reading will be recorded after application of adhesive in similar manner
* Mean increase in denture retention strength will be calculated by subtracting denture retention strength without adhesive from denture retentive strength with adhesive for both study products
* The scores calculated will be filled in Performa (annexure-A)
* The obtained data will be then used to compare diff form of commercially availble denture adhesives (pastes, powder and cushion) for their mean increase in retention strength.
* Then patient will be instructed about how to apply denture adhesives (based on manufacturer' instructions)
* The patient will fill out two attributed questionnaires, before and 1 week after using the denture adhesive. In the questionnaire the satisfaction rating will be determined using valid questionnaires with seven evaluation items: general satisfaction, ability to speak, ease of cleaning, stability, retention, comfort and mastication performance (VAS? Likert scale?)
* The quantitative variable, age of the patients and retention strength was presented as mean+- SD. The qualitative varaible like sex was presented as frequency and percentages. T-test was used to determine the existence if difference of mean retention strength b/w the two form of denture adhesives.
* Data were analyzed using ANOVA and Chi-square tests in SPSS software version 25 software (SPSS version 25.0, SPSS Inc; Chicago, IL, USA) (P<.05)

The score calculated will be filled in the performa (Annexure-A)

ELIGIBILITY:
Inclusion Criteria:

* edentulous patient willing to undergo new complete denture treatments and willing to visit the clinic for denture adjustment as a recall patient
* Healing period of at least 2 months after extraction.

Exclusion Criteria:

* Difficulty responding to questionnaire
* Use of metallic base denture
* Xerostomia
* Ill-fitting dentures
* Neuromuscular disorder
* Smoking habits
* Debilitating diseases
* Immunocompromised
* Maxillofacial defects
* Use a tissue conditioner

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2022-08-18 (Actual); Primary Completion 2023-08-17 (Actual); Study Completion 2023-08-17 (Actual)

PRIMARY OUTCOMES:
To assess the retentive strength of various adhesives on various types of residual ridges using Spring scale | 1 year
  To compare the retentive strengths of different form of commercially available dentures adhesives

SECONDARY OUTCOMES:
To evaluate the effect of various denture adhesives on efficiency of complete denture in patient with different alveolar ridges using a well structured questionnaire | 1 year
  To evaluate the effect of various denture adhesives on efficiency of complete denture in patient with different alveolar ridges using a well structured questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Altamash Institute of dental medicine, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ahmed N, Abbasi MS, Salahuddin A, Tariq L, Siraj S, Das G, Suleman G, Vohra F, Heboyan A. Comparative Analysis of Adhesive Retention and Denture Weight in Different Residual Ridge Morphologies: A Cross-Over Randomized-Controlled Trial. Clin Exp Dent Res. 2025 Feb;11(1):e70118. doi: 10.1002/cre2.70118. PMID 40127129